CLINICAL TRIAL: NCT03807037
Title: Safety of Tocotrienols in Atrial Fibrillation After Coronary Artery Bypass Grafting Surgery: A Randomized Controlled Exploratory Trial
Brief Title: Safety and Efficacy of Tocotrienols in Post-CABG Atrial Fibrillation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Collaborators: Institut Jantung Negara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: T3-AF 34963
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation,tocotrienol,coronary artery bypass grafting
MeSH Terms: conditions — Atrial Fibrillation | interventions — Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Mixed tocotrienols 200mg, twice daily (400mg/day)
  Interventions: Dietary Supplement: Tocotrienols
- Control (Placebo Comparator): Matching Placebo (Placebo oral capsule)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: Tocotrienols — Mixed tocotrienols (derived from palm oil) to be orally administered at 200mg (1 capsule) twice daily, to achieve dosage of 400mg/day
  Other Names: Tocovid Suprabio
  Arms: Treatment
Drug: Placebo oral capsule — Matching placebo to be administered orally at 1 capsule, twice daily
  Arms: Control

SUMMARY:
This study is a prospective, randomized, controlled trial with parallel groups to assess the effects of tocotrienol in the occurrence of atrial fibrillation (AF) post-CABG.

DETAILED DESCRIPTION:
At present, guidelines exist in Europe and the USA on the pharmacological prophylaxis and management of postoperative AF. However, these are subject to a number of limitations including treatment failure, toxicity and pro-arrhythmogenicity. Hence, efforts have been made to develop alternative preventive strategies. The understanding of the role of oxidative stress as a mechanism for AF development has made way for antioxidant vitamins as novel therapeutic and preventive agents.

In view of emerging evidence on the HMG-CoA reductase inhibitory role in the incidence of AF and established inhibitory properties of tocotrienols, we postulate that supplementation with tocotrienols may exert therapeutic advantage in the safety endpoints of post-CABG. The modulation of oxidative stress status and anti-inflammatory via HMG-CoA reductase inhibition may work synergistically in affecting the incidence of AF post-CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females
2. More than 18 years of age
3. Elective, on-pump surgery of coronary artery revascularization, isolated or combined valve surgery

Exclusion Criteria:

1. Less than 18 years of age
2. Refusal to have surgery
3. Urgent or emergency surgery
4. Off-pump surgery
5. Poor LV (EF < 30%)
6. Inability to give informed consent
7. Documented allergy to palm oil or Vitamin E
8. Documented AF or any form of arrhythmia pre-operatively
9. Currently on or indicated for long-term corticosteroid treatment
10. Patients who have been included in any other clinical trial within the previous three months
11. Patients who are on supplementation of Vitamin E or other potent anti-oxidants up to 1 month before randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of AF | 24-48 hours post-operation, up to 6-weeks after discharge
  Between group incidence of post-operative AF

SECONDARY OUTCOMES:
Length of hospital stay (LoHS) after surgery | Up to 2 months post-operation
  1. Total Intensive/coronary care unit length of stay,
  2. Total days of High Dependency Unit stay;
  3. Total hospital length of stay
Health-related quality of life (HRQoL) | 6-weeks after discharge
  Short-Form 36 Questionnaires (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Farouk Musa, MD, Principal Investigator — Monash University Malaysia
Locations (1):
- Institut Jantung Negara, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Musa AF, Dillon J, Taib MEM, Yunus AM, Sanusi AR, Nordin MN, Smith JA. Incidence and Outcomes of Postoperative Atrial Fibrillation after Coronary Artery Bypass Grafting of a Randomized Controlled Trial: A Blinded End-of-cycle Analysis. Rev Cardiovasc Med. 2022 Apr 1;23(4):122. doi: 10.31083/j.rcm2304122. eCollection 2022 Apr. PMID 39076222
- [Derived] Musa AF, Dillon J, Md Taib ME, Yunus AM, Sanusi AR, Nordin MN, Smith JA. A double-blind randomised controlled trial on the effect of Tocovid, a tocotrienol-rich capsule on postoperative atrial fibrillation at the National Heart Institute, Kuala Lumpur: an interim blinded analysis. J Cardiothorac Surg. 2021 Nov 24;16(1):340. doi: 10.1186/s13019-021-01721-6. PMID 34819126